CLINICAL TRIAL: NCT05512182
Title: An Open Label, Single-Arm, Multi-Center Phase II Study to Evaluate the Efficacy of Triplet Combination With Pembrolizumab, Neratinib, and Paclitaxel as a Second Line Treatment in Recurrent/Advanced Gastric Cancer Having Somatic Human Epidermal Growth Factor Receptor Family (EGFR, HER2, HER3, HER4) Mutations or HER2 Amplification/Overexpression
Brief Title: Efficacy of Triplet Combination With Pembrolizumab, Neratinib, and Paclitaxel as a Second Line Treatment in Recurrent/Advanced Gastric Cancer Having Somatic Human Epidermal Growth Factor Receptor Family (EGFR, HER2, HER3, HER4) Mutations or HER2 Amplification/Overexpression
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-1119
Record Dates: First submitted 2022-08-10; First posted 2022-08-23 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Recurrent/Advanced Gastric Cancer
MeSH Terms: conditions — Recurrence | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy (Experimental)
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Pembrolizumab : 200mg/Q3W/IV infusion/Day 1of each 3-week cycle Neratinib : Week 1: 120 mg, Week 2: 160 mg, Week 3 and onwards: 240 mg/QD/Oral/Once daily Paclitaxel : 175mg/m2 /Q3W/IV infusion/Day 1of each 3-week cycle

SUMMARY:
Clinical Indication : HER mutated or HER2 Amplification/Overexpression in Gastric Cancer, 2nd-line Trial Type : Interventional, Open label Treatment Groups : Single arm: Pembrolizumab 200 mg every 3 weeks (Q3W), neratinib at 240 mg once daily (QD), and paclitaxel 175 mg/m2 every 3 weeks (Q3W) Number of trial participants : Approximately 68 patients will be enrolled (with 10% drop-out).

Estimated enrollment period : 24 months Estimated duration of trial : It is estimated that the trial will require approximately 30 months from the time the first patient signs the informed consent until the last patient's last visit.

* First Patient In: Mar 2021
* Last Patient In: Feb 2023
* Last Patient Last Visit: Aug 2023 Duration of Participation : 30 months

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent for the trial.
2. Is male or female at least 19 years of age on the day of signing informed consent.
3. Has a histologically or cytologically confirmed diagnosis of advanced or metastatic gastric adenocarcinoma (systemic metastasis or locally advanced unresectable gastric cancer). A subject must have previously received 1st line chemotherapy using fluoropyrimidine- or platinum-based regimen and showed progression.
4. Has tumors with known activating EGFR, ERBB2, ERBB3, ERBB4 mutations or HER2 amplification by NGS, or HER2 overexpression by IHC or SISH/FISH
5. Has a life expectancy of at least 3 months.
6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
7. Have measurable or evaluable disease determined by RECIST 1.1.
8. Is able to swallow and retain orally administered medication.
9. Have adequate organ function as defined in the following table:

   * white blood cells ≥3000/mm3 and neutrophils ≥1000/mm3
   * platelets ≥100 000/µL
   * hemoglobin ≥9.0 g/dL or ≥5.6 mmol/L
   * AST (SGOT) and ALT (SGPT) ≤3.0 × upper limit of normal (ULN) of the study site (or ≤5.0 × ULN in patients with liver metastases)
   * total bilirubin ≤2.0 × ULN
   * creatinine ≤1.5 × ULN or creatinine clearance >60 mL/min (either measured value or estimated value using the Cockcroft-Gault equation)
10. Has failed in trastuzumab treatment for HER2-positive patients during 1st-line treatment or trastuzumab-naïve for HER2-negative patients measured by IHC or SISH/FISH.
11. Has left ventricular ejection fraction (LVEF) ≥50% measured by multiple-gated acquisition scan (MUGA) or echocardiogram (ECHO).
12. A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 6 months after the last dose of study treatment and refrain from donating sperm during this period.
13. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3; OR
    2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 6 months after the last dose of study treatment.

Exclusion Criteria:

1. Have received second line or more of anticancer treatment (not including adjuvant chemotherapy).
2. Have multiple cancers (with the exception of completely resected basal cell carcinoma, thyroid cancer, stage I squamous cell carcinoma, carcinoma in situ, intramucosal carcinoma, and superficial bladder cancer, and any other cancers that have not recurred for at least 5 years).
3. Have history of hypersensitivity to anti-HER2, immune-oncology drugs.
4. Have brain or leptomeningeal metastases. Patients may be enrolled for the study if they are asymptomatic and require no treatment.
5. Have a tumor with an activating KRAS co-mutation.
6. Have a history of uncontrollable or significant cardiovascular disease meeting any of the following:

   * myocardial infarction within 180 days before study enrolment
   * uncontrollable angina pectoris within 180 days before study enrollment
   * New York Heart Association (NYHA) Class III or IV congestive heart failure
   * uncontrollable hypertension despite appropriate treatment (e.g., systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥90 mmHg lasting 24 hours or more) arrhythmia requiring treatment.
7. Have active, unresolved systemic infection requiring treatment.
8. Are contraindicated for pembrolizumab, neratinib, or paclitaxel, or have severe hypersensitivity (≥Grade 3) to any of those drugs and/or their excipients.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
10. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
11. Have undergone surgery (any surgery involving general anesthesia) within 28 days before study treatment.
12. Have received radiotherapy for gastric cancer within 14 days before study treatment.
13. Have received systemic chemotherapy within 14 days before study treatment.
14. Have received biologic therapy ≤2 weeks or 5 half-lives (t1/2) of the agent used, whichever is shorter, prior to the start of treatment.
15. Have a positive test result for human immunodeficiency virus-1 (HIV-1) antibody.
16. Have hepatitis B surface protein (HBs) antigen and HBV titer >2000 IU/ml (10,000 copy/ml), or hepatitis C virus (HCV) antibody positive result.
17. Are pregnant or breastfeeding, or possibly pregnant.
18. Have any unresolved ≥Grade 2 toxicity (per CTCAE v5.0) from previous anti-cancer therapy at the time of enrollment such as neuropathy, except for alopecia.
19. Are incapable of providing consent for specific reasons, such as concurrent dementia or unwilling for any reason to give consent or to comply with procedures/requirements of this protocol.
20. Are otherwise inappropriate for this study in the investigator's or sub-investigator's opinion.
21. Demonstrates a QTc interval >450 ms for men or >470 ms for women, or has known history of congenital QT-prolongation or Torsade de pointes (TdP).
22. Have significant chronic gastrointestinal disorder with diarrhea as a major symptom (e.g., Crohn's disease, malabsorption, or ≥Grade 2 diarrhea [per CTCAE v5.0] of any etiology at baseline).

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 2 years
  • To determine the objective response rate (ORR) as a second line treatment in recurrent/advanced gastric cancer with somatic HER2 mutations with or without HER2 amplification/overexpression.

SECONDARY OUTCOMES:
overall survival (OS) | 2 years
  overall survival (OS).
progression-free survival (PFS) | 2 years
  according to RECIST 1.1.
disease control rate (DCR) | 2 years
  according to RECIST 1.1.
duration of response (DoR) | 2 years
  duration of response (DoR) according to RECIST 1.1.
Number of participants with treatment-related adverse events as assessed by CTCAE v 5.0 | 2 years
  • To evaluate the safety of pembrolizumab in combination with neratinib and paclitaxel.

CONTACTS AND LOCATIONS:
Overall Officials: SUN YOUNG RHA, Principal Investigator — Yonsei Cancer Center, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No